CLINICAL TRIAL: NCT03708861
Title: Pharmacokinetics of Maraviroc and Boosted Atazanavir Dual Regimen in Stable HIV-infected Patients
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Giovanni Di Perri, Professor, University of Turin, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MARAT; 2014-004692-22 (EudraCT Number)
Record Dates: First submitted 2018-10-14; First posted 2018-10-17 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2019-04

CONDITIONS: HIV Infection
Keywords: maraviroc; atazanavir; ritonavir
MeSH Terms: conditions — HIV Infections | interventions — Maraviroc; Atazanavir Sulfate; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MVC + ATV/r (Experimental): maraviroc (300 mg tablet, 300 mg per day every 24 hours) + atazanavir/ritonavir (300 and 200 mg capsule, 300 and 200 mg per day every 24 hours / 100 mg capsule, 100 mg per day every 24 hours)
  Interventions: Drug: maraviroc (300 mg QD) + atazanavir/ritonavir (300 and 200 mg /100 mg QD)

INTERVENTIONS:
Drug: maraviroc (300 mg QD) + atazanavir/ritonavir (300 and 200 mg /100 mg QD) — Phase 1: switch from tenofovir disoproxil fumarate/emtricitabine (200/245 mg QD)+ atazanavir/ritonavir (300 /100 mg QD) to maraviroc (300 mg QD) + atazanavir/ritonavir (300 /100 mg QD).
  Phase 2: switch from maraviroc (300 mg QD) + atazanavir/ritonavir (300 /100 mg QD) to maraviroc (300 mg QD) + atazanavir/ritonavir (200 /100 mg QD)
  Other Names: CELSENTRI; REYATAZ; NORVIR

SUMMARY:
The purpose of this study is to describe pharmacokinetics of maraviroc (MVC) 300 mg and atazanavir/ritonavir (ATV/r) 200/100 mg QD in HIV-infected stable patients.

DETAILED DESCRIPTION:
The rational of this study is to save therapeutic options, toxicity and costs. The available literature shows that antiretroviral regimens that do not include a nucleoside backbone of tenofovir resulted in less bone and kidney toxicity. Atazanavir dosing 200/100 mg qd represents a simplification strategy correlated with virologic efficacy and a reduction of parameters toxicity associated. Maraviroc is suggested as a possible drug associated to PI/r in dual therapies. Even in this case, the available evidence supports the choice of the dosage of 300 mg/day.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years;
* confirmed HIV-antibodies positivity;
* signed informed consent;
* HIV-RNA <20 cp/ml for the last 24 months;
* no virological failures to PI regimens;
* no major PI resistance associated mutations;
* genotypic tropism for CCR5 co-receptor.

Exclusion Criteria:

* active opportunistic infections or neoplasms;
* need for drugs with known drug-drug interactions with included drugs;
* liver cirrhosis;
* any evidence of tropism for CXCR4 or dual infection;
* pregnancy;
* self-reported adherence<90%;
* HBsAg positivity;
* detectable HCV RNA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
maraviroc (300 mg, QD) + atazanavir/ritonavir (200/100 mg, QD) pharmacokinetic evaluation | within the first 16 weeks after switch
  Number of participants with maraviroc Ctrough>50ng/ml

SECONDARY OUTCOMES:
viral suppression evaluation | week 60
  Number of participants with HIV-RNA<20 cp/ml
CD4 count evaluation | week 60
  Changes in CD4+ count
bone density evaluation | week 60
  Changes in bone mineral density (DEXA femur and spine)
bone metabolism markers evaluation | week 60
  Changes in bone metabolism markers (bALP and vitamin D, PTH)
glomerular and tubular renal function evaluation | week 60
  Changes in proteinuria, glycosuria, phosphaturia and GFR;
lipid metabolism markers evaluation | week 60
  changes in total, HDL, LDL cholesterol and triglycerides
bilirubin evaluation | week 60
  changes in total bilirubin levels

CONTACTS AND LOCATIONS:
Locations (1):
- University of Torino, Torino, Italy

IPD SHARING:
Plan to Share IPD: Undecided